CLINICAL TRIAL: NCT07392775
Title: A Community-Based Approach for ALDH2 Genetic Testing in East Asian Americans
Brief Title: ALDH2 Genetic Testing in East Asian Community
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Jennifer Young, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00222224; 1K01HL173859-01 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult; Flushing
Keywords: East Asian; Alcohol Flushing; ALDH2; ADH1B; Esophageal Cancer; Genetic Testing; Alzheimer's Disease; Cardiovascular Disease
MeSH Terms: conditions — Flushing; Esophageal Neoplasms; Alzheimer Disease; Cardiovascular Diseases | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Flushing Education Only (Active Comparator)
  Interventions: Behavioral: Alcohol Flushing Education
- Alcohol Flushing Education AND Genetic Testing (Experimental)
  Interventions: Behavioral: Genetic Test Results Return; Behavioral: Alcohol Flushing Education

INTERVENTIONS:
Behavioral: Genetic Test Results Return — Returning genetic test results for alcohol flushing genes (i.e., ALDH2, ADH1B)
  Arms: Alcohol Flushing Education AND Genetic Testing
Behavioral: Alcohol Flushing Education — Administering alcohol flushing educational module.

SUMMARY:
The goal of this clinical trial is to learn whether education plus genetic testing for ALDH2*2 and ADH1B*2 is feasible and acceptable and whether it influences modifiable health behaviors in East Asian American adults who experience alcohol flushing when they drink alcohol or have a family history of flushing. The main questions it aims to answer are:

1. Is providing education plus ALDH2*2/ADH1B*2 genetic testing feasible and acceptable in a clinical care context?
2. Does receiving genetic testing results plus education lead to changes in modifiable health behaviors compared with education alone? Researchers will compare education plus genetic testing (intervention arm) to education only (control arm) to see if adding genetic testing improves feasibility/acceptability and supports health behavior change.

Participants will:

1. Complete an education module about alcohol flushing and ALDH2/ADH1B
2. Be randomized to either: (A) Receive genetic testing for ALDH2*2 and ADH1B*2 with results disclosure, or (B) Receive education only.
3. Complete follow-up measures about feasibility, acceptability, and modifiable health behaviors

DETAILED DESCRIPTION:
Alcohol flushing syndrome affects an estimated >500 million individuals worldwide and is strongly associated with functional variants in alcohol metabolism genes, particularly ALDH2 (e.g., ALDH2*2) and ADH1B (e.g., ADH1B*2). ALDH2*2 reduces aldehyde dehydrogenase activity, contributing to acetaldehyde accumulation and is associated with increased risk for alcohol-related morbidity, including certain cancers and cardiometabolic outcomes. Despite the public health relevance, ALDH2/ADH1B implementation in clinical care remains limited, and evidence-based strategies are needed to support equitable and ethical adoption, especially for populations underrepresented in genomics research. This study will engage the East Asian American community to evaluate implementation strategies for ALDH2*2 and ADH1B*2 genetic testing and education in clinical settings and to examine the behavioral impact of returning genetic risk information. Using a pragmatic, randomized comparative effectiveness pilot design, East Asian American adults who self-report alcohol flushing and/or a family history of flushing will be randomized to either: (1) education plus ALDH2*2/ADH1B*2 genetic testing with genotype-informed result disclosure, or (2) education alone. Primary outcomes are feasibility and acceptability of the testing-and-education approach; secondary outcomes include changes in modifiable health behaviors (e.g., alcohol-related decision-making) following education with or without genetic result return. Findings will inform scalable implementation pathways and contribute to equitable integration of genomic testing into routine care for populations experiencing healthcare disparities.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Self-identified as East Asian and/or East Asian American
3. Flush when they drink alcohol or have a family member who flushes when they drink
4. Able to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Alcohol Flushing Genetic Testing in Primary Care | From enrollment to the end of data collection at 8 weeks.
  Feasibility of Intervention Measure (FIM) will be administered to primary care clinicians to measure the extent to which alcohol flushing genetic testing can be successfully used or carried out within a primary care setting. Post-intervention, we will quantitatively assess feasibility of ALDH2 education and genetic testing via 1 questionnaire (4 items total): Feasibility of Intervention Measure (FIM). This 4-item psychometrically-validated measure captures the extent to which individuals believe an implementation strategy is feasible.

SECONDARY OUTCOMES:
Acceptability of Alcohol Flushing Genetic Testing in Primary Care | From enrollment to the end of data collection at 8 weeks.
  Acceptability of Intervention Measure (AIM) assess how agreeable, palatable, or satisfactory alcohol flushing genetic testing is to primary care clinicians. Post-intervention, we will quantitatively assess acceptability of ALDH2 education and genetic testing via 1 questionnaire (4 items total): Acceptability of Intervention Measure (AIM). This 4-item psychometrically-validated measure captures the extent to which individuals believe an implementation strategy is acceptable.
Change(s) in Alcohol Consumption | Alcohol consumption outcome measurements at baseline and one month after educational modules are shared AND after genetic testing results are received.
  Alcohol consumption outcome measurements at baseline and one month after educational modules are shared AND after genetic testing results are received. This results in 3 alcohol outcome measurements total for both arms of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Young, PhD, Principal Investigator — Northwestern U
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Consent language approved by IRB board did not include broad data sharing AND IDP may be identifiable.

REFERENCES:
- [Background] Zhang LL, Wang YQ, Fu B, Zhao SL, Kui Y. Aldehyde dehydrogenase 2 (ALDH2) polymorphism gene and coronary artery disease risk: a meta-analysis. Genet Mol Res. 2015 Dec 28;14(4):18503-14. doi: 10.4238/2015.December.23.38. PMID 26782498
- [Background] Yasue H, Mizuno Y, Harada E. Association of East Asian Variant Aldehyde Dehydrogenase 2 Genotype (ALDH2*2*) with Coronary Spasm and Acute Myocardial Infarction. Adv Exp Med Biol. 2019;1193:121-134. doi: 10.1007/978-981-13-6260-6_7. PMID 31368101
- [Background] Xu YL, Hu YY, Li JW, Zhou L, Li L, Niu YM. Aldehyde dehydrogenase 2 rs671G>A polymorphism and ischemic stroke risk in Chinese population: a meta-analysis. Neuropsychiatr Dis Treat. 2019 Apr 23;15:1015-1029. doi: 10.2147/NDT.S196175. eCollection 2019. PMID 31114208
- [Background] Ding JH, Li SP, Cao HX, Wu JZ, Gao CM, Liu YT, Zhou JN, Chang J, Yao GH. Alcohol dehydrogenase-2 and aldehyde dehydrogenase-2 genotypes, alcohol drinking and the risk for esophageal cancer in a Chinese population. J Hum Genet. 2010 Feb;55(2):97-102. doi: 10.1038/jhg.2009.129. Epub 2009 Dec 11. PMID 20010786
- [Background] Chen J, Huang W, Cheng CH, Zhou L, Jiang GB, Hu YY. Association Between Aldehyde dehydrogenase-2 Polymorphisms and Risk of Alzheimer's Disease and Parkinson's Disease: A Meta-Analysis Based on 5,315 Individuals. Front Neurol. 2019 Mar 28;10:290. doi: 10.3389/fneur.2019.00290. eCollection 2019. PMID 30984100
- See also: Related Info — https://sites.northwestern.edu/younglab/aldh2/